CLINICAL TRIAL: NCT00312728
Title: A Phase II Trial of Bevacizumab in Combination With First- or Second-Line Therapy in Subjects With Treated Brain Metastases Due to Non-Squamous Non-Small Cell Lung Cancer
Brief Title: A Study of Bevacizumab in Combination With First- or Second-Line Therapy in Subjects With Treated Brain Metastases Due to Non-Squamous NSCLC (PASSPORT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVF3752g
Record Dates: First submitted 2006-04-07; First posted 2006-04-11 (Estimated); Results first posted 2011-06-22 (Estimated); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Non-Small Cell Lung Cancer; Brain Neoplasms
Keywords: Brain Cancer; Brain Metastases; Avastin; NSCLC; Lung Cancer; PASSPORT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms; Lung Neoplasms | interventions — Bevacizumab

ARMS (1):
- bevacizumab (Experimental)
  Interventions: Drug: bevacizumab; Drug: First-Line Chemotherapy Agents; Drug: Second-Line Chemotherapy Agents

INTERVENTIONS:
Drug: bevacizumab — 15 mg/kg intravenously (IV) on the first day of each 21- to 28-day cycle (± 4 days); the interval between infusions could not be < 17 days, but could extend beyond 28 days if chemotherapy was delayed to allow recovery from toxicity.
  Other Names: Avastin
Drug: First-Line Chemotherapy Agents — Carboplatin, cisplatin, paclitaxel, docetaxel, gemcitabine, vinorelbine, pemetrexed, or erlotinib administered on Day 1 of every 21-day cycle except gemcitabine, which was administered on Days 1 and 8 of every cycle. Agents were administered as a platinum doublet, or erlotinib alone, at the investigator's discretion. Chemotherapy was administered for a total of 6 planned cycles (up to 8 cycles with prior approval from the Medical Monitor), followed by single-agent bevacizumab therapy. The chemotherapy regimen was to be consistent throughout the study. Erlotinib was administered orally daily.
  All agents were dosed and administered per institutional standards using the respective package insert as a guideline.
Drug: Second-Line Chemotherapy Agents — Erlotinib, pemetrexed, docetaxel, or chemotherapy at the investigator's discretion. Erlotinib was administered orally daily; pemetrexed and docetaxel were administered IV on Day 1 of every 21-day cycle. Single-agent bevacizumab therapy could be continued at the investigator's discretion if the second-line agent was discontinued.
  All agents were dosed and administered per institutional standards using the respective package insert as a guideline.

SUMMARY:
This was an open-label, multicenter, single-arm, Phase II trial of bevacizumab combined with first- or second-line therapy in patients with metastatic non-squamous non-small cell lung cancer (NSCLC) with previously treated central nervous system (CNS) metastases. A total of 115 patients enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Histologically or cytologically confirmed NSCLC except for squamous cell carcinoma
* Treated brain metastases without evidence of progression or hemorrhage after treatment, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period
* Appropriateness for first- or second-line systemic therapy for advanced NSCLC
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Age ≥ 18 years
* For women of childbearing potential and sexually active males, use of an accepted and effective method of contraception (e.g., hormonal or barrier methods, abstinence) prior to study entry and for the duration of the study

Exclusion Criteria:

* Brain biopsy/neurosurgical procedure performed within 3 months prior to Day 1
* Progressive neurologic symptoms
* Active malignancy other than lung cancer
* Current, recent, or planned participation in an experimental drug study
* Prior treatment with an investigational or marketed agent that acts by anti-angiogenesis mechanisms
* Gross hemoptysis within 3 months prior to Day 1
* Inadequately controlled hypertension
* Unstable angina or New York Heart Association Grade II or greater congestive heart failure (CHF)
* Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 1
* Myocardial infarction within 6 months prior to Day 1
* Stroke within 6 months prior to Day 1
* Active symptomatic peripheral vascular disease within 6 months prior to Day 1
* History of significant vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Known hypersensitivity to any components of bevacizumab
* Inadequate organ function
* Serious non-healing wound, ulcer, or bone fracture
* Urine protein/creatinine (UPC) ratio of ≥ 1.0
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1, or anticipation of need for major surgical procedure during the course of the study
* Pregnancy or lactation
* Known evidence of disseminated intravascular coagulation (DIC)
* Active infection or fever > 38.5°C within 3 days prior to Day 1
* Any other medical condition (including mental illness or substance abuse) deemed by the clinician to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Karlin, M.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 110 subjects were to be enrolled at approximately 40 sites to obtain 100 bevacizumab-treated evaluable subjects. Study started 28 NOV 2005 and completed 5 JUN 2009.
Pre-assignment Details: This was an open-label, multicenter, single-arm, Phase II trial of bevacizumab combined with first- or second-line therapy in subjects with metastatic non-squamous non-small cell lung cancer (NSCLC) with previously treated CNS metastases.
Groups:
- Bevacizumab: 15 mg/kg IV on the first day of each 21- to 28-day cycle (+/-4 days) in combination with first or second-line therapy
Period: Overall Study
Arm/Group | Bevacizumab
Started | 115
Completed | 5
Not Completed | 110
Not completed — Progressive disease | 53
Not completed — Adverse Event | 32
Not completed — Withdrawal by Subject | 10
Not completed — Required non-protocol cancer treatment | 2
Not completed — Protocol Violation | 2
Not completed — Other | 10
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab
Number analyzed (Participants) | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (10.6)
Age, Customized [Number; unit: patients]
  18-40 years | 6
  41-64 years | 77
  >=65 years | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 62

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Symptomatic National Cancer Institute's Common Terminology Criteria for Adverse Events v3.0 (NCI CTCAE) Grade ≥2 Central Nervous System (CNS) Hemorrhage
Description: The percentage of participants with symptomatic NCI CTCAE Grade ≥ 2 CNS hemorrhage, defined as the presence of clinical symptoms determined by the investigator to be directly referable to a Grade ≥ 2 CNS hemorrhage.
  Grade 1: Asymptomatic, radiographic findings only Grade 2: Medical intervention indicated Grade 3: Ventriculostomy, intracranial pressure (ICP) monitoring, intraventricular thrombolysis, or operative intervention indicated Grade 4: Life-threatening consequences; neurologic deficit or disability Grade 5: Death
Time Frame: From the first administration of bevacizumab until 60 days after discontinuation of bevacizumab treatment was reported (up to 2 years)
Population: The safety-evaluable population consisted of all patients who received at least one dose of bevacizumab.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 106
percentage of participants | 0 [0 to 2.5]

2. Secondary Outcome: Overall Survival (OS) in First-line Setting
Description: To assess overall survival in the subset of subjects treated in the first-line setting with bevacizumab plus either chemotherapy or erlotinib for non-squamous NSCLC with previously treated brain metastases.
Time Frame: Time from enrollment to death from any cause (up to 2 years)
Population: The first-line efficacy-evaluable population consisted of 70 patients who received at least one dose of bevacizumab.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 70
Months | 11.8 [9.6 to 13.9]

3. Secondary Outcome: Number of Participants With Overall Survival (OS) in First-line Setting [1-Year or More Survival]
Description: Number of Participants with overall survival in the subset of subjects treated in the first-line setting with bevacizumab plus either chemotherapy or erlotinib for non-squamous NSCLC with previously treated brain metastases.
Time Frame: Time from enrollment to death from any cause (up to 2 years)
Population: The first-line efficacy-evaluable population consisted of 70 patients who received at least one dose of bevacizumab.
Measure: Number; unit: participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 70
participants | 30

4. Secondary Outcome: OS in First-line and Second-line Settings
Description: as for outcome 2
Time Frame: Time from enrollment to death from any cause (up to 2 years)
Population: The efficacy-evaluable population consisted of all patients who received at least one dose of bevacizumab.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 106
Months | 12.1 [10.3 to 14.9]

5. Secondary Outcome: Number of Participants With OS in First-line and Second-line Settings [1-Year or More Survival]
Description: To assess the number of participants with overall survival in the subset of subjects treated in the first-line setting with bevacizumab plus either chemotherapy or erlotinib for non-squamous NSCLC with previously treated brain metastases.
Time Frame: Time from enrollment to death from any cause (up to 2 years)
Population: The efficacy-evaluable population consisted of all patients who received at least one dose of bevacizumab.
Measure: Number; unit: participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 106
participants | 49

6. Secondary Outcome: Number of Participants With Selected Adverse Events
Description: Number of participants with selected adverse events (all grades based on NCI CTCAE) included any grade CNS hemorrhage, any grade pulmonary hemorrhage, any grade gastrointestinal (GI) perforation, Grade ≥ 2 arterial thromboembolic event, Grade ≥ 2 left ventricular systolic dysfunction, Grade ≥ 3 non-CNS non-pulmonary hemorrhage, Grade ≥ 3 proteinuria, Grade ≥ 3 proteinuria, Grade ≥ 3 hypertension, any serious adverse event*, and any adverse event leading to study treatment discontinuation.
  *For serious adverse events, please see Adverse Event Reporting Section.
Time Frame: From start of bevacizumab treatment to 60 days following discontinuation of bevacizumab (up to 2 years)
Population: The safety-evaluable population consisted of all patients who received at least one dose of bevacizumab.
Measure: Number; unit: participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 106
participants
  Any grade CNS hemorrhage | 0
  Any grade pulmonary hemorrhage | 4
  Grade ≥ 2 arterial thromboembolic event | 1
  Grade ≥ 3 non-CNS non-pulmonary hemorrhage | 2
  Grade ≥ 3 venous thromboembolic event | 7
  Any grade gastrointestinal perforation | 0
  Grade ≥ 3 hypertension | 3
  Grade ≥ 3 proteinuria | 0
  Grade ≥ 2 left ventricular systolic dysfunction | 0
  Reversible Posterior Leukoencephalopathy Syndrome | 1
  Any event leading to treatment discontinuation | 30

ADVERSE EVENTS:
Time Frame: From start of bevacizumab treatment to 60 days following discontinuation of bevacizumab (up to 2 years).
Arm/Group | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 45/106
Other Adverse Events (participants affected / at risk) | 7/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=106)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 6
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Convulsion (Nervous system disorders) | 4
Ataxia (Nervous system disorders) | 1
BRAIN OEDEMA (Nervous system disorders) | 1
Cerebral Arteriosclerosis (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Leukoencephalopathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient Ischemic Attack (Nervous system disorders) | 1
Pneumonia (Infections and infestations) | 3
Urinary Tract Infection (Infections and infestations) | 2
Diverticulitis (Infections and infestations) | 1
Lobar Pneumonia (Infections and infestations) | 1
Perirectal Abscess (Infections and infestations) | 1
Rectal Abscess (Infections and infestations) | 1
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Chest Pain (General disorders) | 2
Death (General disorders) | 1
Pyrexia (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Failure to Thrive (Metabolism and nutrition disorders) | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1
Mental Status Changes (Psychiatric disorders) | 2
Hypotension (Vascular disorders) | 1
Orthostatic Hypotension (Vascular disorders) | 1
Venous Thrombosis Limb (Vascular disorders) | 1
Hypoaldosteronism (Endocrine disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal Failure Acute (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=106)
Thrombocytopenia (Blood and lymphatic system disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.